CLINICAL TRIAL: NCT04222881
Title: End-to-side Versus Side-to-side Anastomosis With Distal Vein Ligation for Arteriovenous Fistula Creation: a Randomized Controlled Study
Brief Title: End-to-side Versus Side-to-side Anastomosis With Distal Vein Ligation for Arteriovenous Fistula Creation
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: R.18.02.24 - 2018/02/04
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Arterio-venous Fistula
Keywords: End to side anastomosis of arteriovenous fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- End To Side: End to Side Anastomosis
  Interventions: Procedure: AVF anastomosis
- Side To Side: Side To Side Anastomosis
  Interventions: Procedure: AVF anastomosis

INTERVENTIONS:
Procedure: AVF anastomosis — Type of arteriovenous anastomosis

SUMMARY:
End-stage renal disease (ESRD) arises from many heterogeneous disease pathways that alter the function and structure of the kidney irreversibly, over months or years.End-stage renal disease (ESRD) arises from many heterogeneous disease pathways that alter the function and structure of the kidney irreversibly, over months or years. Haemodialysis (HD) is a lifeline therapy for patients with ESRD. Our study to compare methods of AVF creation, side to side and end to side . This randomized controlled trial .

DETAILED DESCRIPTION:
End-to-side versus side-to-side anastomosis with distal vein ligation for arteriovenous fistula creation: A prospective randomized controlled study

Introduction: Arteriovenous fistula (AVF) is the lifeline for patients with chronic renal failure on hemodialysis. The international guidelines recommend patient's referral for access replacement 6 months prior to predicted hemodialysis. The sites being preferred for access replacement are distal arm AVF, proximal arm AVF, basilic vein transposition or graft insertion, respectively (1) Meticulous preoperative assessment and patient selection play great role in achieving functioning AVF with long term patency. AVF maintenance always requires multi-disciplinary approach, with surgeons, nephrologist, dialysis nurses and the patients themselves working hand in hand. Any break in this circle will lead to failure of the AVF, and consequently, failure of hemodialysis. Surgical technique is of paramount importance for long term patency of AVF. There is an ongoing debate about the best technique to do the anastomosis between the artery and the vein; end to side, or side to side. This issue was addressed by very few randomized controlled studies (2,3,4).

Aim of the study: To compare the results of both surgical techniques for creation of arteriovenous anastomosis; End vein to side artery (ETS) versus Side vein to side artery (STS).

Patients and Methods

* Study location: Study protocol will be submitted for approval by Mansoura medical research ethics committee, faculty of medicine, Mansoura University.
* Study design: This is Prospective Randomized controlled trials that is going to be conducted at in department of vascular surgery Mansoura University Hospitals
* Time of study: The study will be conducted during the year 2017-2019.
* Study population: Study population will be on Patients referred to Vascular surgery department for creation of Hemodialysis access. Patients will be advised to undergo elective surgery for AVF once their renal Glomerular Filtration Rate Estimated (eGFR) is less than 15 ml/min.
* Inclusion criteria: All renal failure patients requiring creation of arm AVF, including distal Radio-cephalic, Ulno-basilic, proximal brachio-cephalic or brachio-basilic configurations
* Exclusion criteria: Revision AVF, Synthetic graft AVF or lower limb AVF, Patients with absent distal pulses and chronic ischemia of the upper limb and Recent cannulation of puncture of the vein within 2 weeks before its use in AVF creation.
* Primary End Point: Primary patency of Arterio-venous Fistula and Functional Maturation, ready fistula for cannulation, vein length at least 10 cm, diameter more than 6 mm, depth not more than 6 mm and ability of the access to deliver a flow rate 350 to 400ml/min and maintain dialysis for 4 hours.
* Secondary End Points: Secondary patency, Complication rate failure of maturation, bleeding, infection, steel syndrome and aneurysmal dilatation at anastomosis site
* Target number for recruitment: 50 patients in each group.
* Pre-operative assessment: All patients will undergo clinical assessment as well as routine duplex scan for marking of artery and a patent vein suitable for creation of AVF, with a minimum vein diameter of 2.5 mm for distal fistula and 3 mm for proximal ones.
* Method of Randomization: Computer based randomization.
* Surgical technique: Patients can have the procedure under general, local anesthetic or regional block according to suitability and patients' preference. Mobilization of the suitable artery and vein, creation of fistula using 6/0 prolene for anastomosis in continuous sutures, either ETS or STS with ligation of the distal end of the vein. Arteriotomy size will range from 7 to 10 mm for proximal AVF and from 12 to 15 mm for distal AVF, according to the size of the artery.
* Sites sharing in the study: Mansoura University Hospital
* Post-operative follow-up: Review in clinic on day 6, week 6, months 3 & 6, Duplex scan for assessment of flow in 6 weeks, 3 and 6 months.

Statistical analysis: The data was analyzed using Statistical Package for the Social Sciences. The Significant difference between the flow rate volume in both groups (continuous variable) will be verified by a two-sample test between the two groups. The data analyzed using Cochrane and ANOVA test. Categorical demographic variables were expressed as a proportion of the population and compared with a two-tailed Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* All renal failure patients requiring creation of arm AVF
* Including distal Radio-cephalic, Ulno-basilic, proximal brachio-cephalic or brachio-basilic configurations

Exclusion Criteria:

* Revision AVF, Synthetic graft AVF or lower limb AVF.
* Patients with absent distal pulses and chronic ischemia of the upper limb.
* Recent cannulation of puncture of the vein within 2 weeks before its use in AVF creation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: • Study population will be on Patients referred to Vascular surgery department for creation of Hemodialysis access. Patients will advised to undergo elective surgery for AVF once their renal Glomerular Filtration Rate Estimated (eGFR) is less than 15 ml/min.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-04 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Functional Maturation of Arterio-venous Fistula | Six Months
  Ready fistula for cannulation , vein length at least 10 cm , diameter more than 6 mm ,depth not more than 6 mm and ability of the access to deliver a flow rate 350 to 400ml/min and maintain dialysis for 4 hours.

SECONDARY OUTCOMES:
Complication rate and failure of maturation | Six Months
  Bleeding, infection, steel syndrome and aneurysmal dilatation at anastomosis site

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura, Al Mansurah, Mansoura University, Egypt